CLINICAL TRIAL: NCT00181142
Title: A Phase 3 Study Comparing the Use of Daclizumab vs Thymoglobulin as Induction Therapy in Lung Transplantation
Brief Title: The Use of Daclizumab and Anti-Thymocyte Globulin in Lung Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBIND 8543; 99-06-30-02
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Patients Active and Listed for Lung Transplantation
Keywords: Induciton therapy, Daclizumab, Thymoglobulin, lung transplantation
MeSH Terms: interventions — Daclizumab

INTERVENTIONS:
Drug: Zenapax

SUMMARY:
The purpose of this study is to compare outcomes in patients undergoing lung transplantation, using 2 different induction therapies. Primary outcome is survival and secondary outcomes include freedom from infection and freedom from rejection.

DETAILED DESCRIPTION:
Acute and chronic allograft rejection are two of the common problems limiting and complicating the utility of lung transplantation. The timing and frequency of acute rejection has been shown to be a significant risk factor for the development of chronic allograft rejection. As an adjunct to standard triple immunosuppressive therapy, induction therapy is thought to decrease the incidence of acute rejection.Daclizumab is an interleukin 2 receptor (IL-2) antagonist which is FDA approved as an immunosuppressive agent. Thymoglobulin is an anti-lymphocyte immunosuppressive agent that has been shown in other solid organ transplant studies to be successful in delaying the first episode of rejection but has not decreased the incidence of Obliterative Bronchiloitis (chronic rejection)in lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients accepted and listed for lung transplantation will be considered for randomization

Exclusion Criteria:

* Patients who demonstrate hemodynamic instability, requiring inotropes for greater than 48 hours prior to transplant
* Severe reperfusion pulmonary edema or primary graft dysfunction requiring FiO2 of > 50% and PEEP > 10 cm for greater than 48 hours prior to transplant
* Preoperative renal insufficiency (CrCl < 50 gm.d or serum creatinine > 2.0)
* Pre-operative panel reactive antibodies PRA
* Preoperative recipient bacterial or fungal colonization
* Preoperative antimicrobial suppressive therapy

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1999-10 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality at 2 years.

SECONDARY OUTCOMES:
1)Freedom from 1st >/= A2 rejection episode and incidence of rejection over the first 2 years post-transplant
2)Freedom from infection

CONTACTS AND LOCATIONS:
Overall Officials: John V Conte, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Hospital, Baltimore, Maryland, United States